CLINICAL TRIAL: NCT04739228
Title: Effects of Guided Written Disclosure Protocol on Psychological Distress and Positive Functioning in Persons With Skin Diseases: a Randomized-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Rome (Other)
Collaborators: IRCSS Istituto Dermopatico dell'Immacolata, Fondazione Luigi Maria Monti (Other)
Responsible Party: Principal Investigator, Luca Iani, Associate Professor, European University of Rome
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GDP_2016
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Psychological Distress; Emotional Stress; Skin Diseases; Disclosure
Keywords: Dermatology; Guided Writing Disclosure Protocol; Psychological Distress; Positive Psychology; Randomized-controlled Trial
MeSH Terms: conditions — Stress, Psychological; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Written Disclosure Protocol Group (Experimental): Guided Written Disclosure Protocol is a short-term psychological intervention that stimulates emotional expression, promotes a cognitive reworking of stressful illness events and facilitates the integration between emotional and cognitive processing of traumatic experiences. Intervention aimed at enhancing patients' quality of life, psychological well-being, and emotional regulation, and reducing psychosocial distress.
  Interventions: Behavioral: Guided Written Disclosure Protocol Group
- Active Control Group (Active Comparator)
  Interventions: Behavioral: Active Control Group

INTERVENTIONS:
Behavioral: Guided Written Disclosure Protocol Group — The writing task consists of three sessions of 20 minutes each, with an interval of one week between each other. In the first session, patients were asked to describe the onset of illness, describing chronologically and detailed places, images, sounds and actions, as they are followed and detached from the emotions. In the second session, the patients were asked to write about thoughts and emotions felt during the illness experience, talking about the impact that illness had on their daily lives and how it had changed their personal attitude to life itself. In the third and final session, the patients were asked to analyze subjective new skills acquired.
  Arms: Guided Written Disclosure Protocol Group
Behavioral: Active Control Group — The writing task also consists of three sessions of 20 minutes each, with an interval of one week between each other. In all three writing sessions, patients were asked to report the daily activities during the last week, without focusing on the emotional aspects.
  Arms: Active Control Group

SUMMARY:
We conducted a randomized-controlled trial of Guided Written Disclosure Protocol for dermatological patients with the aim of reducing psychological distress, expressive suppression, and skin-related symptoms, and improving spiritual well-being, cognitive reappraisal, and sense of coherence.

DETAILED DESCRIPTION:
Sample size assessment: A recent meta-analysis reported a study which showed that Guided Written Disclosure Protocol reach on effect size of 0.89 on psychosocial outcomes (Gidron et al., 2002; Mogk et al., 2006). Power analysis showed that with an alpha of 0.05 and a power of 0.80, we needed a sample of 34 participants to detect effect sizes of 0.89 and higher.

Plan for missing data: Occasional missing values were imputed by calculating, for each participant, the average score for each subscale and then replaced.

Statistical analysis plan: We conducted a 2 (group) X 2 (time [pre-treatment vs. post-treatment]) repeated measures multivariate analysis of variance (MANOVA) for a set of variables.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Diagnosis of psoriasis or systemic sclerosis by a board-certified dermatologist.

Exclusion Criteria:

* Patients with certified mental disorders (e.g., psychotic illness, major depressive disorder)
* Patients undergoing psychotherapy for at least 6 months in the last 3 years;
* Patients who currently receive psychopharmacological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Pre-test to Post-test and Follow-up in Spiritual Well-Being, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-Test (before the intervention), Post-Test (30 days after the baseline assessment)
  Spiritual well-being will be measured with the FACIT-Sp (minimum value=0; maximum value=48, with higher scores indicating a better outcome), a questionnaire assessing faith, peace and meaning
Change from Pre-test to Post-test and Follow-up in Psychological Distress, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-Test (before the intervention), Post-Test (30 days after the baseline assessment)
  Psychological distress will be measured with the GHQ-12 (minimum value=1; maximum value=4, with higher score indicating greater outcome).

SECONDARY OUTCOMES:
Change from Pre-test to Post-test and Follow-up in Emotion Regulation, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-Test (before the intervention), Post-Test (30 days after the baseline assessment)
  Emotion regulation will be measured with ERQ (minimum value=1; maximum value=7), a questionnaire assessing expressive suppression and cognitive reappraisal.
Change from Pre-test to Post-test and Follow-up in Skin-related Quality of Life, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-Test (before the intervention), Post-Test (30 days after the baseline assessment)
  Skin-related Quality of Life will be measured with Skindex 29 (minimum value=1; maximum value=5, with higher score indicating a worse outcome), a questionnaire assessing symptoms, emotions, and functioning.
Change from Pre-test to Post-test and Follow-up in Sense of Coherence, which will be reported in the outcome measure results data table as means and standard deviations. | Pre-Test (before the intervention), Post-Test (30 days after the baseline assessment)
  Sense of Coherence will be measured with SOC-13 (minimum value=1; maximum value=7, with higher score indicating a greater outcome), a questionnaire assessing comprehensibility and meaningfulness of human experience

CONTACTS AND LOCATIONS:
Overall Officials: Luca Iani, PhD, Principal Investigator — European University of Rome
Locations (1):
- IRCSS Istituto Dermopatico dell'Immacolata, Fondazione Luigi Maria Monti, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol
Time Frame: Data will become available after the study will be published
Access Criteria: Through the depository Figshare

REFERENCES:
- [Result] Gidron Y, Duncan E, Lazar A, Biderman A, Tandeter H, Shvartzman P. Effects of guided written disclosure of stressful experiences on clinic visits and symptoms in frequent clinic attenders. Fam Pract. 2002 Apr;19(2):161-6. doi: 10.1093/fampra/19.2.161. PMID 11906981
- [Result] Mogk C, Otte S, Reinhold-Hurley B, Kroner-Herwig B. Health effects of expressive writing on stressful or traumatic experiences - a meta-analysis. Psychosoc Med. 2006 Nov 16;3:Doc06. PMID 19742069